CLINICAL TRIAL: NCT01633567
Title: A Culturally Targeted and Individually Tailored Smoking Cessation Intervention for LGBT Smokers
Brief Title: Culturally Targeted & Individually Tailored Smoking Cessation Study: LGBT Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Cancer Institute (NCI) (NIH); Howard Brown Health Center (Other)
Responsible Party: Principal Investigator, Alicia Matthews, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0538; R01DA023935 (NIH)
Record Dates: First submitted 2012-05-30; First posted 2012-07-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cigarette Smoking
Keywords: Smoking Cessation; Cigarette Smoking; Tobacco; LGBT; LGBTQ
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Culturally Targeted Cessation Program (Experimental): The culturally targeted program will include the same cognitive and behavioral approaches and smoking education content that is used in the standard program. As such, we will maintain the integrity of the core program. However, cultural targeting of that program has been informed by local LGBT focus group input and testing, the available literature on LGBT smoking rates and behaviors, feedback from a panel of LGBT health experts, and data collected as part of a previous study.
  Interventions: Behavioral: Culturally Targeted Cessation Program
- Non-Targeted Cessation Program (Active Comparator): Non-culturally targeted program with cognitive and behavioral approaches and smoking education content.
  Interventions: Behavioral: Non-Targeted Cessation Program

INTERVENTIONS:
Behavioral: Culturally Targeted Cessation Program — The culturally targeted version of the behavioral counseling intervention will consist of six group-based smoking cessation counseling sessions. Each smoking cessation therapy session will last approximately 90 minutes and will begin two weeks before the quit date. In addition, participants will be provided nicotine replacement therapy and peer support sessions will occur between the group sessions.
  Arms: Culturally Targeted Cessation Program
Behavioral: Non-Targeted Cessation Program — Behavioral counseling intervention will consist of six group-based smoking cessation counseling sessions. Each smoking cessation therapy session will last approximately 90 minutes and will begin two weeks before the quit date. In addition, participants will be provided nicotine replacement therapy and peer support sessions will occur between the group sessions.
  Arms: Non-Targeted Cessation Program

SUMMARY:
For the approximately 4.6 million LGBT persons in the U.S., smoking rates among those living in urban areas are roughly twice that of heterosexuals. Targeted interventions have shown great promise in reducing health risk behaviors across a variety of behaviors and population groups by enhancing the relevance of the health information. The primary aim of this study is to test the efficacy of a culturally targeted group-based smoking cessation intervention (vs. a non-targeted intervention) on smoking outcomes among lesbian, gay, bisexual, and transgender (LGBT) smokers. The investigators anticipate that the culturally targeted intervention will be more effective at helping LGBT smokers to successfully stop smoking than will the non-targeted intervention.

DETAILED DESCRIPTION:
In Phase 1 of this study we used focus groups to establish the cultural appropriateness and acceptability of the targeted elements of the intervention for the LGBT population. For Phase 2 of this study, we seek to enroll 400 participants in a randomized controlled trial of the targeted intervention vs. a non-targeted, comparison condition. Both conditions will consist of group counseling sessions combined with nicotine replacement therapy and peer support. We expect that quit rates, stage of readiness, perceived benefits, self-efficacy, and treatment adherence will be higher among those who received the targeted intervention than those in the non-targeted intervention. Furthermore, we expect that a stronger LGBT cultural identification and salience of that identity will be associated with more satisfaction and adherence to the targeted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self identify as lesbian, gay, bisexual, or transgender
* Age 18-65
* Current cigarette smoker
* Desire to quit smoking (self-report rating of interest in quitting)
* Relatively healthy, with no medical conditions that would adversely interact with study parameters (see exclusion criteria for specific details)
* Agree to attend behavioral counseling sessions, be randomized, and be followed-up
* Agrees to use nicotine patch and has no prior adverse reactions to patch
* Has stable residence and telephone and can provide the name of an outside household collateral family member or close friend for contact and follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
7-Day Point Prevalence Smoking Quit Rates 1 Month Post Quit Date | Assessed 1 month after quit date
  7-Day point prevalence smoking quit rates will serve as the main outcome measure and will be obtained from Time Line Follow-Back (TLFB) interviews.
7-Day Point Prevalence Smoking Quit Rates 3 Months Post Quit Date | Assessed 3 months after quit date
  7-Day point prevalence smoking quit rates will serve as the main outcome measure and will be obtained from Time Line Follow-Back (TLFB) interviews.
7-Day Point Prevalence Smoking Quit Rates 6 Months Post Quit Date | Assessed 6 months after quit date
  7-Day point prevalence smoking quit rates will serve as the main outcome measure and will be obtained from Time Line Follow-Back (TLFB) interviews.
7-Day Point Prevalence Smoking Quit Rates 12 Months Post Quit Date | Assessed 12 months after quit date
  7-Day point prevalence smoking quit rates will serve as the main outcome measure and will be obtained from Time Line Follow-Back (TLFB) interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia K Matthews, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Howard Brown Health Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matthews AK, McConnell EA, Li CC, Vargas MC, King A. Design of a comparative effectiveness evaluation of a culturally tailored versus standard community-based smoking cessation treatment program for LGBT smokers. BMC Psychol. 2014 May 30;2(1):12. doi: 10.1186/2050-7283-2-12. eCollection 2014. PMID 25566383
- See also: Research Partner Agency — http://www.howardbrown.org
- See also: University of Illinois at Chicago Website — http://www.uic.edu